CLINICAL TRIAL: NCT06099054
Title: Ultrasound-guided Pigtail Catheter Versus Intercostal Tube Drainage of Non-traumatic Exudative Pleural Effusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Hassan Sayed, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pigtail versus ICT
Record Dates: First submitted 2023-09-22; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Pleural Effusion
Keywords: pigtail versus intercostal tube
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to either group:
  Group I (Intervention group): in which pleural effusion will be drained using pigtail catheter under US guidance.
  Group II (Control group): in which pleural effusion will be drained using ICT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pigtail group (Experimental): composed of 40 patients in which pleural effusion will be drained using pigtail catheter under US guidance
  Interventions: Device: Pigtail catheter
- ICT group (Active Comparator): composed of 40 patients in which pleural effusion will be drained using ICT
  Interventions: Device: Intercostal tube

INTERVENTIONS:
Device: Pigtail catheter — Pigtail catheter will be inserted using Seldinger technique under US guidance to drainage exudative pleural effusion by a trained radiologist
  Arms: pigtail group
Device: Intercostal tube — Chest tube will be inserted according to BTS guideline for insertion of ICT by a trained thoracic surgeon
  Arms: ICT group

SUMMARY:
Primary Aims:

To compare the performance of pigtail catheter to that of ICT in drainage of pleural effusion of medical aetiology regarding:

1. Various complications(mainly wound pain) that result from either therapeutic approach.
2. Success of complete drainage.
3. Compare the duration needed for complete drainage.

Secondary Aims:

To evaluate both techniques in terms of:

1. Degree of patient's mobility that either technique permits.
2. Percentage of patients that can be managed on outpatient settings by either approach

DETAILED DESCRIPTION:
The pleural cavity is a space between the visceral and parietal pleura that contains a subtle amount of serous fluid (10 to 20ml) this fluid act as a lubricant to the pleural surface for proper gliding during respiration . Accumulation of abnormal amount of pleural fluid occurs under various pathological disorders, each of which manifests with a different physical and biochemical characteristics of the effused pleural fluid, it may be serous,pus,blood,or chyle.

Long standing undrained accumulated pleural fluid can lead to serious complications: like lung collapse leading to respiratory failure, fibrosis or scarring of the pleural membranes and underlying lung tissue, empyema, septic shock and even death in severe circumstance .

So we always seek to drain accumulated pleural fluid; Chest tubes connected to underwater seal have largely replaced open thoracotomy and rib resection in draining exudative pleural effusion and are now considered the standard method . However Intercostal tube drainage poses risks and hazards: large size of the tube that make it more painful more tissue destructive with more injury to intercostal arteries and nerves, the incisional insertion is also painful and results in more tissue dissection, moreover the tube is heavy as it need water seal to work so causing patient discomfort and increase liability of slippage.

Recently pigtail catheter has been employed to drain accumulated pleural fluid .pigtail catheter has many advantages: it has small caliber , which makes it less painful, less tissue destruction, less Injurious to intercostal nerves and vessels, Additionally it has a suction power with unidirectional valve which abolishes the need for underwater seal; thus avoiding the heavy weight of bottles and decreasing the risk of accidental slippage, inserted with trocar under ultrasonographic guidance decreasing liability of lung injury.

Previous studies compared pigtail versus chest tube in drainage of pleural effusion show .A total of 92 patients were included in the study, 57 (61.9%) patients in pigtail group and 35 (31.8%) in ICD group. Causes of pleural effusion included were pneumonia, malignancy,TB. the study had revealed that pigtail catheter had higher success rate less painful with no significant difference at mean duration of drainage..At other study data collected retrospectively from 60 patient aged more than 18 year 30 patients had an intercostal chest tube and 30 patients had pigtail catheters found that no statistically significant difference between pigtail and ICT at success rate and duration of drainage but pigtail found less painful with less incidence of complication regarding pneumothorax and catheter kinking and slippage .

However these studies have some limations first study was observational study not randomised, second study was retrospective with small sample size. Both studies have no clear definitions of outcomes , not focus on complications mainly wound pain as primary outcome and didn't answer the question of recurrence or drainage failure of pleural effusion after pigtail catheter drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Non-traumatic non-iatrogenic exudative pleural effusion necessitating drainage.
3. Loculated pleural effusion where positive colour doppler sign is preserved

Exclusion Criteria:

1. Traumatic or iatrogenic pleural effusion.
2. Transudative pleural effusion (subjected to treatment of the underlying cause and diuretic therapy).
3. Exudative pleural effusion amenable for medical treatment
4. Large-volume, easily accessible, free non-loculated empyema.
5. Pleural infections with loculated pleural effusion but showing negative colour doppler sign.
6. Malignant pleural effusion with potentially inexpnasible underlying lung (thick pleural peel, central airway obstruction), life expectancy < 1 month or asymptomatic.
7. Patients with uncorrected bleeding tendency (INR > 1.5, Platelet count < 50.000/mm3).
8. Inability or refusal to sign written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
1) Degree of Pain/discomfort elicited by the Intervention: | 10 day
  The visual analogue Scale from 0 TO 10 will be used to score reported pain or discomfort
2) Adverse outcomes complicating either line of intervention | through study completion, an average of 1 year
  (e.g., new onset pneumothorax or haemothorax, subcutaneous emphysema, fluid leakage around the wound, organ puncture, re-expansion pulmonary oedema, pneumonia, blockade of the drain, kinking or malposition).
3) Success of Complete Drainage | through study completion, an average of 1 year
  Number of patients with complete drainage:
  Complete drainage will be considered if all the following conditions are met:
  Amount of drained fluid < 50 cc of serous/ hemo-serous fluid (no pus or gross bleeding) for two successive days.
  No accompanying air leak in the previous 12 hours. Radiological resolution (no residual free pleural fluid seen by chest US and lung expansion against chest wall as detected by chest US and CXR)
4) Duration needed for Complete Drainage: | 15 day
  Duration (in days) will be counted from the day of drain insertion to the day of drain removal

SECONDARY OUTCOMES:
5) Degree of Patient's Mobility: | 0ne week
  A modification of a 6-item survey assessing the patient's sense of security with a chest drain will be used. Patients are to be asked to report:
  1. How confident they are moving with the chest drain without limitation in activities.
  2. How confident they are moving with the chest drain without concerns about accidental slippage/removal of the drainage set.
  3. How confident they are moving with the chest drain without concerns about accidental damage/breakage to the drainage set.
  Patients are to report their answer to this question on a 5-point Likert's scale, where 5 meant "definitely yes" and 1 meant "definitely not".
6) Duration of Hospital stay. | "through study completion, an average of 1 year
  number of patients need hospitalization and duration they will spend at hospital
7) Number of Patients Managed on Outpatient Settings. | "through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hossam El-din Galal, Prof.Dr, Principal Investigator — Assiut Univeristy; Hamdy Mohammad Ibrahim, lecturer, Study Director — Assiut Univeristy; Sara Mohammed Hashem, lecturer, Study Director — Assiut Univeristy

REFERENCES:
- [Background] Chubb SP, Williams RA. Biochemical Analysis of Pleural Fluid and Ascites. Clin Biochem Rev. 2018 May;39(2):39-50. PMID 30473591
- [Background] Karkhanis VS, Joshi JM. Pleural effusion: diagnosis, treatment, and management. Open Access Emerg Med. 2012 Jun 22;4:31-52. doi: 10.2147/OAEM.S29942. eCollection 2012. PMID 27147861
- [Background] Broaddus VC, Light RW. Pleural effusion. In:Broaddus VC, Ernst JD, King TE, et al, eds. Murray and Nadel's Textbook of Respiratory Medicine. 7th ed. Philadelphia, PA: Elsevier; 2022:chapater108
- [Background] Monaghan SF, Swan KG. Tube thoracostomy: the struggle to the "standard of care". Ann Thorac Surg. 2008 Dec;86(6):2019-22. doi: 10.1016/j.athoracsur.2008.08.006. PMID 19022041
- [Background] Munnell ER. Thoracic drainage. Ann Thorac Surg. 1997 May;63(5):1497-502. doi: 10.1016/s0003-4975(97)00082-9. PMID 9146363
- [Background] Liu YH, Lin YC, Liang SJ, Tu CY, Chen CH, Chen HJ, Chen W, Shih CM, Hsu WH. Ultrasound-guided pigtail catheters for drainage of various pleural diseases. Am J Emerg Med. 2010 Oct;28(8):915-21. doi: 10.1016/j.ajem.2009.04.041. Epub 2010 Feb 25. PMID 20825924
- [Background] Gammie JS, Banks MC, Fuhrman CR, Pham SM, Griffith BP, Keenan RJ, Luketich JD. The pigtail catheter for pleural drainage: a less invasive alternative to tube thoracostomy. JSLS. 1999 Jan-Mar;3(1):57-61. PMID 10323171
- [Background] Khare R*, Anand K, Agrawal P, Yadav A. Comparative analysis of pigtail catheter versus intercostal tube drainage for pleural effusion: a tertiary centre study. Khare R et al. Int Surg J. 2023 Jan;10(1):105-109
- [Background] Mathis G. Pleura. In: Mathis G, ed. Chest sonography. 3rd ed. Heidelberg: Springer-Verlag, 2011;30-32
- [Background] Yang PC, Luh KT, Chang DB, Wu HD, Yu CJ, Kuo SH. Value of sonography in determining the nature of pleural effusion: analysis of 320 cases. AJR Am J Roentgenol. 1992 Jul;159(1):29-33. doi: 10.2214/ajr.159.1.1609716.
- [Background] Reuß J., "Sonographic imaging of the pleura: Nearly 30 years experience," European Journal of Ultrasound, vol. 3, no. 2, pp. 125-139, 1996.
- [Background] SELDINGER SI. Catheter replacement of the needle in percutaneous arteriography; a new technique. Acta Radiol (Stockh). 1953 May;39(5):368-76. doi: 10.3109/00016925309136722. No abstract available. PMID 13057644
- [Background] Laws D, Neville E, Duffy J; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the insertion of a chest drain. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii53-9. doi: 10.1136/thorax.58.suppl_2.ii53. No abstract available. PMID 12728150
- [Background] Fox V, Gould D, Davies N, Owen S. Patients' experiences of having an underwater seal chest drain: a replication study. J Clin Nurs. 1999 Nov;8(6):684-92. doi: 10.1046/j.1365-2702.1999.00307.x. PMID 10827615